CLINICAL TRIAL: NCT02636543
Title: Evaluation of the Information Letter to Relatives in the Context of Genetic Assessments
Acronym: LIPEG
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/32
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Transmission of Information to the Relatives After Genetic Diagnosis
Keywords: genetic diagnosis; information; letter model

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 2a-patient: 75 patients who attended a genetic counselling consultation.
  Interventions: Other: Questionnaire after the reading of letter B.
- Group 2a-public: 75 persons belonging to general population.
  Interventions: Other: Questionnaire after the reading of letter B.
- Group 2b-patient: 75 patients who attended a genetic counselling consultation (those patients are different than patients from group 2a-).
  Interventions: Other: Questionnaire after the reading of letter B.; Other: Questionnaire after the reading of letters A and B
- Group 2b-public: 75 persons belonging to general population (those persons are different than patients from group 2a).
  Interventions: Other: Questionnaire after the reading of letter B.; Other: Questionnaire after the reading of letters A and B
- Group 2b-professional: 75 genetic professionals.
  Interventions: Other: Questionnaire after the reading of letter B.; Other: Questionnaire after the reading of letters A and B

INTERVENTIONS:
Other: Questionnaire after the reading of letter B. — Oral questionnaire after the reading of letter B.
Other: Questionnaire after the reading of letters A and B — Oral questionnaire after the reading of letters A and B during individual interview.
  Groups: Group 2b-patient; Group 2b-professional; Group 2b-public

SUMMARY:
The decree of June 20th 2013 (n° 2013-527) suggests a protocol regarding the transmission of information to the relatives after genetic diagnosis of a serious condition. This decree includes a specific model of letter that can be sent to relatives by genetic professionals. We evaluated the understanding and feelings after the reading of the decree's letter (letter A) on patients and the public. A focus group drafted a new version of the letter (letter B) through these observations. The two letter models (A vs B) are compared in terms of impact through precise items (understanding and feelings) on three populations: patients, public and genetic professionals. Assumption is made that the letter B will be preferred to the letter A. Overall, we aim at giving a letter formulation accommodating as many people as possible to standardize practices.

DETAILED DESCRIPTION:
The recent publication of the decree of June 20th 2013 (n° 2013-527) suggests a protocol regarding the transmission of information of the relatives after genetic diagnosis of a serious condition allowing preventative or care measures. In the case a mutation career refuses to directly inform other members of his family, option is to call on services of a genetic professional for the transmission of its family information. This decree includes a specific model of letter that can be sent to relatives by genetic professionals.

The main objective of the present study is the standardization of the procedure concerning the information to relatives by all genetic professionals. It would allow the same format of information in all families involved.

The first part (study 1a) evaluated the understanding and feelings after the reading of the decree's letter (letter A) on patients and the public, through the use of an individual and oral questionnaire. Interviews with the patients, public, genetic professionals and people who have received this letter completed the study 1a (study 1b). A focus group (accounting different genetic professionals and patient associations) composed a new version of letter (letter B) through these observations (study 1c).

The second part will compare the two letters model (A vs B) impact through precise items on three populations: patients, public and genetic professionals. This study will allow to:

* Evaluate how the letter composed by the focus group (letter A) is understood and perceived by the patients and the public with the same methodology as study 1a (study 2a) ;
* Compare the two letters model (A vs B) to describing the preference of patients, public and genetic professionals (study 2b).

The expected results would help us to choose the letter accommodating as many people as possible to standardize practices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* French native speaker
* informed person
* person whose non-opposition has been received
* public: person who never attended a genetic counselling consultation
* professional: geneticist and genetic counsellors working in France

Exclusion Criteria:

* study 2a : person who took part of study 2b
* study 2b : person who took part of study 2a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 2a-patient: 75 patients who attended a genetic counselling consultation.
  * Group 2a-public: 75 persons belonging to the general population who never attended genetic counselling consultation.
  * Group 2b-patient: 75 patients who attended a genetic counselling consultation.
  * Group 2b-public: 75 persons belonging to general population who never attendeda genetic counselling consultation. These persons are different than persons from group 2a-person.
  * Group 2b-professionnal: 75 genetic professionals (geneticist and genetic counsellor).
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Score of understanding questionnaire after reading letter B. | 1 day
Proportion of persons who prefer the letter B. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Cécile ZORDAN, Ms, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - University Hospital Bordeaux, Bordeaux, Aquitaine
  - Hôpital Universitaire de Strasbourg, Strasbourg, Aquitaine
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Rennes - Hôpital SUD, Rennes
  - CHU de Toulouse - Hôpital Purpan, Toulouse